CLINICAL TRIAL: NCT01343069
Title: Safety Analysis in Regard to the Introduction of Surgical Checklists in the Operation Rooms in a Tertiary Care Center
Brief Title: Safety Improvement and Checklist Application
Acronym: SICA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient quality of data
Sponsor: Regional Hospital of Bolzano (Other)
Responsible Party: Principal Investigator, Matthias Bock, Safety Analysis in Regard to the Introduction of Surgical Checklists in the Operation Rooms in a Tertiary Care Center, Regional Hospital of Bolzano
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: check4outcome2
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Complications; Outcome
Keywords: safety; team; team performance; surgery; outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- before surgical checklist (No Intervention)
- after implementation surgical checklist (Active Comparator)
  Interventions: Procedure: implementation surgical checklist

INTERVENTIONS:
Procedure: implementation surgical checklist — a checklist according to the suggestions raised by the WHO is implementated
  Arms: after implementation surgical checklist

SUMMARY:
The study investigates the impact of the introduction of a surgical checklist on the incidence of complications and mortality within 30 days after surgery in patients scheduled for elective non-cardiac surgery. Patients scheduled for elective surgical procedures lasting longer than 20 minutes at are eligible. Surgery is performed in a single tertiary care center. Study design is an open trial before and after intervention (implementation of the checklist "safe surgery saves lifes").

ELIGIBILITY:
Inclusion Criteria:

* elective surgery in general or regional anesthesia lasting > 15 min

Exclusion Criteria:

* urgent surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
number of complications after elective surgery | within 30 days
  comparison of number of complications in the two study arms before and after introduction of the checklist

SECONDARY OUTCOMES:
mortality | 30 days
  evaluation of 30-days mortality

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Bock, MD, Study Director — Central Hospital Bolzano Italy